CLINICAL TRIAL: NCT04569838
Title: A Multicenter, Single-arm Phase II Study to Evaluate the Efficacy and Safety of Bendamustine Hydrochloride Injection in Subjects With Rituximab-resistant Indolent B-Cell Non-Hodgkin's Lymphomas
Brief Title: A Study to Evaluate the Efficacy and Safety of Bendamustine Hydrochloride Injection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BDMS-C10IICS-PRT
Record Dates: First submitted 2020-09-25; First posted 2020-09-30 (Actual); Last update posted 2020-09-30 (Actual); Status verified 2020-09

CONDITIONS: Indolent B-Cell Non-Hodgkin's Lymphomas
MeSH Terms: interventions — Bendamustine Hydrochloride

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bendamustine hydrochloride injection (Experimental): Bendamustine hydrochloride injection 120 mg/m² or 100 mg/m² intravenously (IV) on Day 1 and Day 2 of 21-day cycle (6-8 cycles maximum) for non-hodgkin's lymphomas or chronic lymphocytic leukemia. After 6-8 cycles, the course of treatment could be added based on patient's benefit and investigator's determination.
  Interventions: Drug: Bendamustine hydrochloride injection

INTERVENTIONS:
Drug: Bendamustine hydrochloride injection — Bendamustine is a bifunctional alkylating agent. It cross-links DNA single strand and double strand by alkylation,then destroys the function and synthesis of DNA, and makes the DNA and protein, protein and protein cross-linking, has potential to treat various tumors

SUMMARY:
This is a study to evaluate the efficacy and safety of Bendamustine Hydrochloride Injection in subjects with Rituximab-resistant Indolent B-Cell Non-Hodgkin's Lymphomas.

ELIGIBILITY:
Inclusion Criteria:

* 1. Inert lymphoma, including follicular lymphoma (FL), extranodal marginal zone B-cell lymphomas of the mucosa-associated lymphoid tissue (MALT), lymphoplasmacytic lymphoma, mantle cell lymphoma, small lymphocyte B-cell lymphoma and chronic lymphoblastic leukemia (CLL).

  2. At least one measurable lesion with the longest diameter > 1.5 cm and the short diameter > 1.0 cm, or the peripheral blood B lymphocyte ≥ 5.0×109/L.

  3.Adequate laboratory indicators. 4. Has received one to three chemotherapy regimens (with or without rituximab) before enrollment.

  5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1; Life expectancy ≥ 3 months.

  6. Understood and signed an informed consent form.

Exclusion Criteria:

* 1. Patients who could not tolerate bendamustine treatment according to the investigators' judgment.

  2. Has received anti-tumor treatment (including major surgery) in the last 4 weeks.

  3. Transformed into high malignant lymphoma (secondary to low-grade follicular lymphoma); grade 3B follicular lymphoma.

  4. Has received corticosteroids regularly in the last 4 weeks. 5. Has a history of central nervous system disease or central nervous system disease.

  6. Has other tumors. 7. Has suffered from serious infection and other drugs or mental illness,which affects signing informed consent form and follow-up visit.

  8. Pregnant or breastfeeding women. 9. Has participated in other clinical trials within three months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2012-05 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate（ORR） | Baseline up to 30 weeks
  Percentage of participants achieving complete response (CR) and partial response (PR).
Duration of Response (DOR) | Baseline up to 30 weeks
  DOR defined as time from earliest date of disease response to earliest date of disease progression based on radiographic assessment.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | Baseline up to 30 weeks
  PFS defined as the time from randomization until the first documented progressive disease (PD) or death from any cause.
Overall Survival (OS) | Baseline up to 30 weeks
  OS defined as the time from randomization to death from any cause. Subjects who do not die at the end of the extended follow-up period, or were lost to follow-up during the study, were censored at the last date they were known to be alive.

CONTACTS AND LOCATIONS:
Locations (11):
- China (11):
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - First People's Hospital of Foshan, Foshan, Guangdong
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Guangzhou First People's Hospital, Guangzhou, Guangdong
  - Southern Medical University Nanfang Hospital, Guangzhou, Guangdong
  - Shenzhen People's Hospital, Shenzhen, Guangdong
  - Guangxi Medical University Affiliated Tumor Hospital, Nanning, Guangxi
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Affiliated Hospital of Nantong University, Nantong, Jiangsu
  - The Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu